CLINICAL TRIAL: NCT02343484
Title: Intradiscal Combination of Gelified Ethanol and Pulsed Radiofrequency Versus Gelified Ethanol Injection for the Treatment of Chronic Discogenic Low Back Pain. A Randomized Controlled Trial.
Brief Title: Intradiscal Gelified Ethanol and Pulsed Radiofrequency Versus Gelified Ethanol Injection for Discogenic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Chrysanthi Batistaki, Assistant Professor of Anesthesiology, 2nd Department of Anesthesiology, School of Medicine, University of Athens, Greece, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2/8-2-13
Record Dates: First submitted 2015-01-13; First posted 2015-01-22 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Low Back Pain
Keywords: pulsed radiofrequency; gelified ethanol
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gelified ethanol (Active Comparator): Gelified ethanol (Discogel) is a sterile, implantable medical solution containing ethyl alcohol, cellulose derivative product and an opaque agent (tungsten). The implant is administered within the affected intervertebral disc nucleus pulposus, via a fine needle which is guided into the center of the disc, transdermally. The implant causes migration of fluid (by hydrophilic and osmotic phenomena) from the periphery towards the center, causing disk reinforcement. Filling of the annulus fibrosus tears interrupts the outflow of inflammatory factors towards dorsal root ganglions, dura and posterior longitudinal ligament.
  Interventions: Drug: Gelified ethanol
- Gelified ethanol combined to pulsed radiofrequency (Active Comparator): Pulsed radiofrequency treatment is performed intradiscally for the management of chronic discogenic low back pain.Intradiscal pulsed radiofrequency is first applied and then combined to gelified ethanol injection via the same radiofrequency needle.
  Interventions: Drug: Gelified ethanol combined to pulsed radiofrequency

INTERVENTIONS:
Drug: Gelified ethanol combined to pulsed radiofrequency — Gelified ethanol (Discogel) is a sterile, implantable medical solution which is administered within the affected intervertebral disc nucleus pulposus, via a fine needle which is guided into the center of the disc, transdermally. Pulsed radiofrequency treatment is performed intradiscally for the management of chronic discogenic low back pain. The intradiscal pulsed radiofrequency is first applied and then combined to gelified ethanol injection via the same radiofrequency needle.
  Other Names: Discogel; PRF
  Arms: Gelified ethanol combined to pulsed radiofrequency
Drug: Gelified ethanol — Gelified ethanol is a sterile, implantable medical solution which is administered within the affected intervertebral disc nucleus pulposus, via a fine needle which is guided into the center of the disc, transdermally.
  Other Names: Discogel
  Arms: Gelified ethanol

SUMMARY:
Many different minimally invasive techniques have been used for the treatment of chronic discogenic low back pain refractory to conservative treatments, with various results. The aim of this study is to assess the efficacy of the combination of intradiscal pulsed radiofrequency and gelified ethanol versus gelified ethanol alone, on pain and quality of life of patients sufferring from chronic discogenic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Discogenic low back pain > 6 months,
* pain refractory to conservative treatment,
* no other aetiology for pain,
* pain reported during provocative discography according to standard criteria,
* MRI imaging indicating disk degenarative disease

Exclusion Criteria:

* Red flags for low back pain,
* lumbosacral radiculopathy,
* extruded or sequestered lumbar disc,
* severe spinal stenosis,
* facet joint syndrome,
* sacroiliac joint pain,
* neurological disorders,
* psychiatric disorders,
* rheumatoid arhtritis, ancylosing spondylitis, other autoimmune arthritis,
* coagulation disorders,
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Rating Scale (NRS) | One, three, six and twelve months after the procedure.
  Mean pain intensity assessed by VAS 1, 3, 6 and 12 months after the procedure.
Change in Rolland Morris questionnaire | One, three, six and twelve months after the procedure.
  Functional status of patient assessed by Rolland Morris questionnaire 1, 3, 6 and 12 months after the procedure.

SECONDARY OUTCOMES:
Change in Quality of life (EQ 5D) | One, three, six and twelve months after the procedure.
  Quality of life assessed via EQ 5D questionnaire 1, 3, 6 and 12 months after the procedure
Change in Satisfaction from therapy ( assessed via NRS 0-10) | One, three, six and twelve months after the procedure.
  Satisfaction from therapy assessed via NRS 0-10 1, 3, 6 and 12 months after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon Hospital, 1 Rimini str., Athens, Greece

REFERENCES:
- [Background] Bellini M, Romano DG, Leonini S, Grazzini I, Tabano C, Ferrara M, Piu P, Monti L, Cerase A. Percutaneous injection of radiopaque gelified ethanol for the treatment of lumbar and cervical intervertebral disk herniations: experience and clinical outcome in 80 patients. AJNR Am J Neuroradiol. 2015 Mar;36(3):600-5. doi: 10.3174/ajnr.A4166. Epub 2014 Nov 13. PMID 25395657
- [Background] Guarnieri G, De Dominicis G, Muto M. Intradiscal and intramuscular injection of discogel((R)) - radiopaque gelified ethanol: pathological evaluation. Neuroradiol J. 2010 Apr;23(2):249-52. doi: 10.1177/197140091002300216. Epub 2010 Apr 20. PMID 24148546
- [Background] Theron J, Guimaraens L, Casasco A, Sola T, Cuellar H, Courtheoux P. Percutaneous treatment of lumbar intervertebral disk hernias with radiopaque gelified ethanol: a preliminary study. J Spinal Disord Tech. 2007 Oct;20(7):526-32. doi: 10.1097/BSD.0b013e318033e860. PMID 17912130
- [Background] Manchikanti L, Abdi S, Atluri S, Benyamin RM, Boswell MV, Buenaventura RM, Bryce DA, Burks PA, Caraway DL, Calodney AK, Cash KA, Christo PJ, Cohen SP, Colson J, Conn A, Cordner H, Coubarous S, Datta S, Deer TR, Diwan S, Falco FJ, Fellows B, Geffert S, Grider JS, Gupta S, Hameed H, Hameed M, Hansen H, Helm S 2nd, Janata JW, Justiz R, Kaye AD, Lee M, Manchikanti KN, McManus CD, Onyewu O, Parr AT, Patel VB, Racz GB, Sehgal N, Sharma ML, Simopoulos TT, Singh V, Smith HS, Snook LT, Swicegood JR, Vallejo R, Ward SP, Wargo BW, Zhu J, Hirsch JA. An update of comprehensive evidence-based guidelines for interventional techniques in chronic spinal pain. Part II: guidance and recommendations. Pain Physician. 2013 Apr;16(2 Suppl):S49-283. PMID 23615883
- [Background] Jung YJ, Lee DG, Cho YW, Ahn SH. Effect of intradiscal monopolar pulsed radiofrequency on chronic discogenic back pain diagnosed by pressure-controlled provocative discography: a one year prospective study. Ann Rehabil Med. 2012 Oct;36(5):648-56. doi: 10.5535/arm.2012.36.5.648. Epub 2012 Oct 31. PMID 23185729
- [Background] Rohof O. Intradiscal pulsed radiofrequency application following provocative discography for the management of degenerative disc disease and concordant pain: a pilot study. Pain Pract. 2012 Jun;12(5):342-9. doi: 10.1111/j.1533-2500.2011.00512.x. Epub 2011 Oct 19. PMID 22008239
- [Background] Fukui S, Rohof O. Results of pulsed radiofrequency technique with two laterally placed electrodes in the annulus in patients with chronic lumbar discogenic pain. J Anesth. 2012 Aug;26(4):606-9. doi: 10.1007/s00540-012-1385-7. Epub 2012 Apr 5. PMID 22476553
- [Background] Fukui S, Nitta K, Iwashita N, Tomie H, Nosaka S, Rohof O. Results of intradiscal pulsed radiofrequency for lumbar discogenic pain: comparison with intradiscal electrothermal therapy. Korean J Pain. 2012 Jul;25(3):155-60. doi: 10.3344/kjp.2012.25.3.155. Epub 2012 Jun 28. PMID 22787545